CLINICAL TRIAL: NCT04435925
Title: Inflammatory Effect Comparison Between Fentanyl and Remifentanil in Mastectomy Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Christopher Ryalino, Principal Investigator, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UNUD-CTR-FK110620-001
Record Dates: First submitted 2020-06-11; First posted 2020-06-17 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Breast Disease; Anesthesia; Inflammatory Response
MeSH Terms: conditions — Breast Diseases | interventions — Remifentanil; Fentanyl

STUDY DESIGN:
Intervention Model Description: This is a single-blind, randomized control trial. It provides a controlled treatment of general anesthesia with an opioid regimen between remifentanil and fentanyl.
Who Masked: Participant
Masking Description: The opioid selection disguised to the patient. Eligible subjects will be randomized so that each research subject has the same opportunity to be included in both groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remifentanil (Active Comparator): Patients assigned to this group will receive IV Remifentanil as an opioid for general anesthesia.
  Interventions: Drug: Remifentanil
- Fentanyl (Placebo Comparator): Patients assigned to this group will receive IV Fentanyl as an opioid for general anesthesia.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Remifentanil — Loading dose: 0.5 mcg/kg Maintenance dose: 1 mcg/kg/minute
  Arms: Remifentanil
Drug: Fentanyl — Loading dose: 2 mcg/kg Maintenance dose: 0.4 mcg/kg/30-minutes
  Arms: Fentanyl

SUMMARY:
Mastectomy triggers stress and inflammation responses due to tissue trauma. Surgical stress will increase levels of hormones (adrenocorticotropic hormone, cortisol, antidiuretic hormone, epinephrine, norepinephrine, and dopamine) and inflammatory cytokines (Tumor Necrotic Factor-α, interleukin-1, interleukin-2, and interleukin-6) in the body. This causes insulin resistance, gluconeogenesis, and glycolysis, and impaired insulin secretion, which results in hyperglycemia due to intraoperative stress. Intraoperative hyperglycemia increases postoperative complications and mortality. Inhibition of hyperglycemia due to operative stress and stress hormones with good anesthetic management in improving patient outcomes.

The choice of opioid type plays an important role in suppressing the perioperative stress and inflammatory response. Opioids are an alternative, besides the use of regional anesthetic techniques which have been proven to suppress the perioperative stress response. Fentanyl is one of the phenylpiperidine synthetic opioids. Large doses of fentanyl can reduce stress responses but also increase side effects, such as hemodynamic instability and decrease T-cell function.

Remifentanil provides unique pharmacokinetic benefits through nonspecific esterase enzyme metabolism, so it has a very fast onset and half-life. In addition, remifentanil also provides benefits in reducing the production of interleukin 6 cytokines (IL-6) and tumor necrosis factor α (TNF-α) and inhibits neutrophil migration through the endothelial layer.

The stress response to stress and inflammation is directly proportional to the dose of remifentanil given. It is reported that remifentanil can suppress cortisol response according to increasing dose.

Winterhalter et al. and Lee et al. reported that remifentanil is better at suppressing the stress response than fentanyl. On the other hand, Bell et al. showed no difference in cortisol and hemodynamic levels between the two groups.

The goal of this study is to see if remifentanil provides less increase in serum epinephrine level, norepinephrine level, platelet to lymphocyte ratio (PLR), lymphocyte to monocyte ratio (LMR), and blood glucose level at one-hour and 24-hours postoperative in patients undergoing mastectomy surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a mastectomy under general anesthesia
* Patients aged 30-65 years old
* ASA physical status: I-II

Exclusion Criteria:

* Refusal to be included in the study
* History of opioid allergies
* Long-term use of steroids
* Patients on β blockers medication
* History of diabetes, autoimmune disease, or heart disease

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Epinephrine | 1-hour (postoperative)
  Serum epinephrine level
Epinephrine | 24-hours (postoperative)
  Serum epinephrine level
Norepinephrine | 1-hour (postoperative)
  Serum norepinephrine level
Norepinephrine | 24-hours (postoperative)
  Serum norepinephrine level
PLR | 1-hour (postoperative)
  platelet-to-lymphocyte ratio
PLR | 24-hours (postoperative)
  platelet-to-lymphocyte ratio
LMR | 1-hour (postoperative)
  lymphocyte-to-monocyte ratio
LMR | 24-hours (postoperative)
  lymphocyte-to-monocyte ratio
Glucose | 1-hour (postoperative)
  serum glucose level
Glucose | 24-hours (postoperative)
  serum glucose level

CONTACTS AND LOCATIONS:
Overall Officials: I Gusti AG Hartawan, Principal Investigator — Udayana University
Locations (1):
- Sanglah General Hospital, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No